CLINICAL TRIAL: NCT03740061
Title: The Evaluation of Acute Sarcopenia in Hospitalized Elderly: Muscle Characteristics Assessment Through Ultrasound
Brief Title: Muscle Assessment Through Ultrasound in the Evaluation of Acute Sarcopenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Hospital Universitario Ramon y Cajal (Other); Universitaire Ziekenhuizen KU Leuven (Other); Medical University of Bialystok (Other); Catholic University of the Sacred Heart (Other); Universitat Autonoma de Barcelona (Other); Jagiellonian University (Other); Universitat Pompeu Fabra (Other); Istanbul University (Other); University of Oldenburg (Other)
Responsible Party: Principal Investigator, Stany Perkisas, Principal investigator, Universiteit Antwerpen
Other Study IDs: SARCUS2
Record Dates: First submitted 2018-10-23; First posted 2018-11-14 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Sarcopenia
Keywords: Ultrasound; Assessment; Acute sarcopenia; Hospitalized older people
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Antwerp
  Interventions: Diagnostic Test: Ultrasonographic assessment of muscle
- Barcelona
  Interventions: Diagnostic Test: Ultrasonographic assessment of muscle
- Istanbul
  Interventions: Diagnostic Test: Ultrasonographic assessment of muscle
- Oldenburg
  Interventions: Diagnostic Test: Ultrasonographic assessment of muscle
- Krakow
  Interventions: Diagnostic Test: Ultrasonographic assessment of muscle
- Bialystok
  Interventions: Diagnostic Test: Ultrasonographic assessment of muscle
- Rome
  Interventions: Diagnostic Test: Ultrasonographic assessment of muscle
- Madrid
  Interventions: Diagnostic Test: Ultrasonographic assessment of muscle
- Leuven
  Interventions: Diagnostic Test: Ultrasonographic assessment of muscle

INTERVENTIONS:
Diagnostic Test: Ultrasonographic assessment of muscle — Ultrasonographic assessment of quadriceps muscle

SUMMARY:
Traditionally, muscle mass - a part of the concept of sarcopenia - is measured by computed tomography (CT) or dual-energy X-ray absorptiometry (DEXA) scan. These devices are not always easily available in clinical practice and cannot be used bedside. An innovation in sarcopenia is the assessment of muscle mass and quality with ultrasound. Because this device is much more available and applicable in all patients, diagnosis of acute sarcopenia would be much easier with ultrasound. Moreover, if other factors that contribute to accelerated decline in muscle mass and function can be determinated, the sensiblisation and early screening for acute sarcopenia in those individuals can hopefully prevent them from declining.

DETAILED DESCRIPTION:
Methods Study design A prospective, multicenter, international observational study will be conducted. The study is designed to determine the effect of hospitalisation due to acute illness on the changes in muscle mass and muscle function. The secondary endpoint of the study is to identify health related parameters associated with the development of acute sarcopenia.

Subjects Inclusion criteria Patients admitted between the 1st of December 2018 until the 31th of November 2019 will be eligible for inclusion. Included wards for admission are: internal medicine, acute geriatrics, orthogeriatrics and rehabilitation. Age limit will be set on 65 years and older.

Exclusion criteria Patients on dialysis will be excluded because of possible metabolic features. Individuals with paresis of the lower limbs or hemiparesis due to a stroke will be excluded because of neurological involvement that can influence the results. Hypo-or hyperthyroid patients will be excluded because of the role of thyroid hormones in muscle homeostasis. Pitting oedema of the legs (due to heart failure, anasarca oedema, renal failure or liver cirrhosis) or severely dehydrated patients will be excluded because fluid shifts could influence the ultrasound measurement results. Because of possible previous changes in muscle mass, architecture and function, patients with systemic connective tissue disorders, myositis, calcification and ossification of muscle, systemic atrophies primarily affecting the central nervous system and demyelinating diseases of the central nervous system will be excluded. Patients using chronic oral corticosteroids will be excluded.

Settings and locations The study will be a multicenter study held in different university and tertiary teaching hospitals throughout Europe.

Measurements

Patient characteristics Date of birth, gender, height and weight will be registered. If the patient is bedridden, weight can be measured through either weight chairs or weight measuring lifts. Height will be estimated using the ulna length or knee height. Date of admission and discharge will be noted. The home care setting of the patient will be registered. The main reason of hospital admission will be registered.

Comorbidities on admission will be registered through the Cumulative Illness Rating Scale for Geriatrics (CIRS-G). The CIRS-G was designed to estimate the survival of elderly persons, assessing disease severity using a score from 0 to 4 in 14 different categories of organ systems: cardiac, vascular, hematological, respiratory, ophthalmological and otorhinolaryngological, upper gastro-intestinal, lower gastro-intestinal, hepatic and pancreatic, renal, genito-urinary, musculoskeletal and tegumental, neurological, endocrine/metabolic/breast and psychiatric. Score '0' stands for 'no problem affecting that system', score '1' stands for 'current mild problem or past significant problem', score '2' stands for 'moderate disability or morbidity', score '3' stands for 'severe problem' and score '4' stands for 'extremely severe problem'.

Laboratory values that will be checked are either nutritional through albumin and prealbumin, inflammatory through C-reactive protein (CRP) and white blood cell count, and the measurement of 25-hydroxyvitamin D (25-OH-vitamin D). Blood samples will be collected on day of admission. Laboratory values that are not expected to fluctuate strongly (albumin, pre-albumin, 25-OH-vitamin D) will be taken within the first 5 days of admission.

Muscle mass In order to obtain reliable and consistent measurements, all ultrasonography will be done by an ultrasonographist that is trained to perform the measurements proposed. For the measurements, a linear probe of 5 cm width will be used. Frequency of the beam will be set on 12 MHz.

Patients should not have had any physical exercise in the 30 minutes before the measurement. Muscles should be completely relaxed and patients should be placed in the supine position, with hips in neutral position and knees fully extended. The dominant leg will be taken for the measurements. To calculate the relative muscle thickness values, the total length of muscle will be noted.

Ultrasonographic data of the four bellies of the quadriceps muscle (rectus femoris, vastus lateralis, vastus medialis, vastus intermedius) will be taken. Measuring points will be specified according to the propositions of the SARCUS-working group. Muscle thickness, fascicle length, pennation angle, muscle cross-sectional area and echo-intensity of all muscles listed will be taken.

The first measurement will be taken as early as possible within 48 hours after admission at the latest. Follow-up measurements will be taken according to the type of ward the patient is admitted to. For patients that are expected to be hospitalized for a limited time (<5 days), the follow-up measurement will be done 3 days after initial measurement. For patients that are expected to be hospitalized for a longer time (>7 days), measurements will be repeated 7 days after initial measurement, to be repeated after another 7 days as long as the patient is hospitalized.

Muscle strength and function Muscle strength will be measured through hand grip strength using a Jamar dynamometer, using the Southampton protocol. The first measurement will be taken as early as possible within 48 hours after admission at the latest. Follow-up measurements will be taken according to the type of ward the patient is admitted to. For patients that are expected to be hospitalized for a limited time (<5 days), the follow-up measurement will be done 3 days after initial measurement. For patients that are expected to be hospitalized for a longer time (>7 days), measurements will be repeated 7 days after initial measurement, to be repeated after another 7 days as long as the patient is hospitalized. Measurement will be done directly after the ultrasonographic assessment. If feasible, muscle function will be measured through gait speed, using the 4-meter walking test at usual gait speed. In case of those bedridden, gait speed will not be measured.

In-hospital activity Registration of activity level during hospitalisation will be performed by means of pedometers in those centers that have access to these devices. Both amount of steps and step length will be noted, and total walked distance per day can hereby be calculated.

Nutritional status Nutritional state of the patient will be registered through the Mini-Nutritional Assessment - Short Form (MNA-SF). For diagnosis of malnutrition, the new Global Leadership Initiative on Malnutrition (GLIM)-criteria will be used.

Questionnaires The SARC-F and FRAIL-scale will be completed as routine screening questionnaires for sarcopenia and frailty, respectively. The SAR-QOL questionnaire will be used to evaluate the self-reported quality of life.

Statistical analysis Databases will be kept up in a Microsoft Access database. Statistical analysis will be done by using SPSS Statistics version 24. Descriptive analyses will be used for determining the clinical and demographic characteristics. A Kolmogorov-Smirnov test will be used to verify the normal distribution of the different variables. Further statistical analyses will be performed by Chi Square test, Fisher exact, Mann-Whitney U test or Fisher exact test, depending on the distribution and the nature of the variables analysed. P-values of ≤0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* All participants ages 65 years AND
* Admitted to one of the ward of one of the centers in the given time period.

Exclusion Criteria:

* Patients on dialysis will be excluded because of possible metabolic features.
* Individuals with paresis of the lower limbs or hemiparesis due to a stroke will be excluded because of neurological involvement that can influence the results.
* Hypo-or hyperthyroid patients will be excluded because of the role of thyroid hormones in muscle homeostasis.
* Pitting oedema of the legs (due to heart failure, anasarca oedema, renal failure or liver cirrhosis) or severely dehydrated patients will be excluded because fluid shifts could influence the ultrasound measurement results.
* Because of possible previous changes in muscle mass, architecture and function, patients with systemic connective tissue disorders, myositis, calcification and ossification of muscle, systemic atrophies primarily affecting the central nervous system and demyelinating diseases of the central nervous system will be excluded.
* Patients using chronic oral corticosteroids will be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All participants ages 65 years or older and admitted to one of the ward of one of the centers in the given time period.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Change over 7 days in ultrasonographic measured muscle thickness (in centimeter) in the four bellies of the quadriceps muscle | 7 days
  Change over 7 days in ultrasonographic measured muscle thickness (in centimeter) in the four bellies of the quadriceps muscle
Change over 7 days in ultrasonographic measured muscle cross-sectional area (in square centimeter) in the four bellies of the quadriceps muscle | 7 days
  Change over 7 days in ultrasonographic measured muscle cross-sectional area (in square centimeter) in the four bellies of the quadriceps muscle
Change over 7 days in ultrasonographic measured muscle pennation angle (in degrees) in the four bellies of the quadriceps muscle | 7 days
  Change over 7 days in ultrasonographic measured muscle pennation angle (in degrees) in the four bellies of the quadriceps muscle
Change over 7 days in ultrasonographic measured muscle fascicle length (in centimeter) in the four bellies of the quadriceps muscle | 7 days
  Change over 7 days in ultrasonographic measured muscle fascicle length (in centimeter) in the four bellies of the quadriceps muscle
Change over 7 days in ultrasonographic measured muscle echo-intensity (gray values in Houndsfield units) in the four bellies of the quadriceps muscle | 7 days
  Change over 7 days in ultrasonographic measured muscle echo-intensity (gray values in Houndsfield units) in the four bellies of the quadriceps muscle

SECONDARY OUTCOMES:
Influence of muscle thickness on muscle strength measured by hand grip strength | 7 days
  Determining what the influence of (changes in) muscle thickness (in centimeter) in the four bellies of the quadriceps muscle is on muscle strength measured by hand grip strength (kg)
Influence of muscle cross-sectional area on muscle strength measured by hand grip strength | 7 days
  Determining what the influence of (changes in) muscle cross-sectional area (in square centimeter) in the four bellies of the quadriceps muscle on muscle strength measured by hand grip strength (kg)
Influence of muscle pennation angle on muscle strength measured by hand grip strength | 7 days
  Determining what the influence of (changes in) muscle pennation angle (in degrees) in the four bellies of the quadriceps muscle is on muscle strength measured by hand grip strength (kg)
Influence of muscle fascicle length on muscle strength measured by hand grip strength (kg) | 7 days
  Determining what the influence of (changes in) muscle fascicle length (in centimeter) in the four bellies of the quadriceps muscle is on muscle strength measured by hand grip strength (kg)
Influence of muscle echo intensity on muscle strength measured by hand grip strength (kg) | 7 days
  Determining what the influence of (changes in) muscle echo intensity (gray values in Houndsfield units) in the four bellies of the quadriceps muscle is on muscle strength measured by hand grip strength (kg)
Influence of muscle thickness on muscle function measured by short physical performance battery | 7 days
  Determining what the relation is between (changes in) muscle thickness (in centimeter) in the four bellies of the quadriceps muscle and muscle function measured by short physical performance battery
Influence of muscle cross-sectional area on muscle function measured by short physical performance battery | 7 days
  Determining what the influence of (changes in) muscle cross-sectional area (in square centimeter) in the four bellies of the quadriceps muscle on muscle function measured by short physical performance battery
Influence of muscle pennation angle on muscle function measured by short physical performance battery | 7 days
  Determining what the influence of (changes in) muscle pennation angle (in degrees) in the four bellies of the quadriceps muscle is on muscle function measured by short physical performance battery
Influence of muscle fascicle length on muscle function measured by short physical performance battery | 7 days
  Determining what the influence of (changes in) muscle fascicle length (in centimeter) in the four bellies of the quadriceps muscle is on muscle function measured by short physical performance battery
Influence of muscle echo intensity on muscle function measured by short physical performance battery | 7 days
  Determining what the influence of (changes in) muscle echo intensity (gray values in Houndsfield units) in the four bellies of the quadriceps muscle is on muscle function measured by short physical performance battery

CONTACTS AND LOCATIONS:
Overall Officials: Stany Perkisas, MD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- ZNA Middelheim, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT03740061/Prot_SAP_000.pdf